CLINICAL TRIAL: NCT00174746
Title: A Placebo- and Active-Controlled (Ciclesonide Metered-Dose Inhaler), Randomized, Parallel-Group, Dose-Range Finding Study of Ciclesonide Administered by Dry Powder Inhaler (Ultrahaler) in Adult and Adolescent Patients With Persistent Asthma
Brief Title: Dose Response Study of Inhaled Ciclesonide (Glucocorticosteroid) to Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI6153
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Asthma
Keywords: Glucocorticosteroid; Dose response; Bronchospasm
MeSH Terms: conditions — Asthma; Bronchial Spasm

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: AVE2635A

SUMMARY:
To investigate the efficacy and safety of ciclesonide inhaled into the lungs in a range of doses in a new dry powder inhaler compared to ciclesonide inhaled into the lungs using a metered dose inhaler

ELIGIBILITY:
Inclusion Criteria:

* Males or females 12 years or older; History of persistent bronchial asthma for at least 6 months; Documented use of an inhaled steroid for at least 1 month before screening; At screening, FEV1 40% or more of predicted normal and at randomization, FEV1 between 40 and 80% predicted normal; Reversibility of FEV1 by at least 12% and 200 ml post-bronchodilator; Be able to use oral inhalers; Non-smokers

Exclusion Criteria:

* History of life-threatening asthma; other pulmonary diseases; URI within 4 weeks before screening; Use of systemic steroids within 1 month before screening or more than 3 times in previous 6 months; beta-adrenergic blocking agent use; More than 2 in-patient hospitalizations or ER visits due to asthma exacerbations in the prior year before screening; Pregnant or breast-feeding females; Females of child-bearing potential not using adequate means of birth control; Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease; Abnormal clinical laboratory parameters that would limit participation in the study or interfere with interpretation of study results; History of drug or alcohol abuse; Treatment with any investigational product within 30 days prior to study entry

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1145 (Actual)
Dates: Start 2005-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Primary endpoint will be the change from baseline to week 6 in FEV1

SECONDARY OUTCOMES:
PK parameters measured after 4 weeks of treatment. Change from baseline in serum cortisol pre-and post ACTH stimulation, AM and PM peak expiratory flow rates, AM and PM asthma symptoms, and albuterol use after 6 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States